CLINICAL TRIAL: NCT03625466
Title: An Exploratory Phase 2, 2-part, Randomized, Double-blind, Placebo-controlled Study With a Long-term, Open-label Period to Explore the Impact of Lumacaftor/Ivacaftor on Disease Progression in Subjects Aged 2 Through 5 Years With Cystic Fibrosis, Homozygous for F508del
Brief Title: A Study to Explore the Impact of Lumacaftor/Ivacaftor on Disease Progression in Subjects Aged 2 Through 5 Years With Cystic Fibrosis, Homozygous for F508del
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX16-809-121; 2017-003761-99 (EudraCT Number)
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Results first posted 2021-12-08 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded in Part 1, and Open label in Part 2
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Placebo (Placebo Comparator): Participants received placebo matched to LUM/IVA in placebo-controlled period for 48 weeks.
  Interventions: Drug: Placebo
- Part 1: LUM/IVA (Experimental): Participants weighing less than (<)14 kilograms (kg) at screening received LUM 100 milligrams (mg)/IVA 125 mg fixed-dose combination (FDC) every 12 hours (q12h) in placebo-controlled period for 48 weeks. Participants weighing greater than or equals to (>=)14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h in placebo-controlled period for 48 weeks.
  Interventions: Drug: LUM/IVA
- Part 2: Overall LUM/IVA (Experimental): Participants who received either placebo or LUM/IVA in placebo-controlled period administered LUM/IVA (either LUM 100 mg/IVA 125 mg FDC q12h or LUM 150 mg/IVA 188 mg FDC q12h as per their body weight for participants <6 years of age at week 48 and LUM 200 mg/IVA 250 mg FDC q12h regardless of their body weight for participants >=6 years of age at week 48) in open-label period for 48 weeks.
  Interventions: Drug: LUM/IVA

INTERVENTIONS:
Drug: LUM/IVA — FDC tablets or granules for oral administration.
  Other Names: Lumacaftor/Ivacaftor; VX-809/VX-770
  Arms: Part 2: Overall LUM/IVA
Drug: LUM/IVA — FDC granules for oral administration.
  Other Names: Lumacaftor/Ivacaftor; VX-809/VX-770
  Arms: Part 1: LUM/IVA
Drug: Placebo — Placebo matched to LUM/IVA for oral administration.
  Arms: Part 1: Placebo

SUMMARY:
This study will explore the impact of lumacaftor/ivacaftor (LUM/IVA) on disease progression in subjects aged 2 through 5 years with cystic fibrosis (CF), homozygous for F508del (F/F).

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with confirmed diagnosis of CF.
* Homozygous for F508del (F/F).
* Subjects who weigh ≥8 kg without shoes and wearing light clothing at the Screening Visit.

Key Exclusion Criteria:

* Any clinically significant laboratory abnormalities at the Screening Visit that would interfere with the study assessments or pose an undue risk for the subject.
* Solid organ or hematological transplantation.
* History of any illness or comorbidity reviewed at the Screening Visit that, in the opinion of the investigator, might confound the results of the study.

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Charite Paediatric Pulmonology Department, Berlin
  - Justus-Leibig-Universitat Zentrum fur Kinderheilkunde und Jugendmedizin, Giessen
  - Hannover Medical School, Hanover
  - Heidelberg Cystic Fibrosis Center, Heidelberg
  - Universitatsklinikum Schleswig-Holstein, Klinik für Kinder- und Jugendmedizin, Lübeck

REFERENCES:
- [Derived] Stahl M, Roehmel J, Eichinger M, Doellinger F, Naehrlich L, Kopp MV, Dittrich AM, Sommerburg O, Ray P, Maniktala A, Xu T, Conner S, Joshi A, Mascia M, Wielputz MO, Mall MA. Long-Term Impact of Lumacaftor/Ivacaftor Treatment on Cystic Fibrosis Disease Progression in Children 2-5 Years of Age Homozygous for F508del-CFTR: A Phase 2, Open-Label Clinical Trial. Ann Am Thorac Soc. 2024 Nov;21(11):1550-1559. doi: 10.1513/AnnalsATS.202402-201OC. PMID 39173175
- [Derived] Stahl M, Roehmel J, Eichinger M, Doellinger F, Naehrlich L, Kopp MV, Dittrich AM, Lee C, Sommerburg O, Tian S, Xu T, Wu P, Joshi A, Ray P, Duncan ME, Wielputz MO, Mall MA. Effects of Lumacaftor/Ivacaftor on Cystic Fibrosis Disease Progression in Children 2 through 5 Years of Age Homozygous for F508del-CFTR: A Phase 2 Placebo-controlled Clinical Trial. Ann Am Thorac Soc. 2023 Aug;20(8):1144-1155. doi: 10.1513/AnnalsATS.202208-684OC. PMID 36943405

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned in 2 parts: Part 1 (Placebo-controlled Period) and Part 2 (Open-label Period). The primary and secondary efficacy analyses were planned for only Part 1.
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF) aged 2 to 5 years.
Period: Placebo-controlled Period (48 Weeks)
Arm/Group | Part 1: Placebo | Part 1: LUM/IVA | Part 2: Overall LUM/IVA
Started | 16 | 35 | 0
Completed | 16 | 33 | 0
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal of Consent (not due to AE) | 0 | 1 | 0
Period: Open-label Period (48 Weeks)
Arm/Group | Part 1: Placebo | Part 1: LUM/IVA | Part 2: Overall LUM/IVA
Started | 0 | 0 | 49
Completed | 0 | 0 | 48
Not Completed | 0 | 0 | 1
Not completed — Withdrawal of Consent (not due to AE) | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants who have received at least 1 dose of study drug.
Groups:
- Part 1: LUM/IVA: Participants weighing <14 kg at screening received LUM 100 mg/IVA 125 mg FDC every q12h in placebo-controlled period for 48 weeks. Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h in placebo-controlled period for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: LUM/IVA | Total
Number analyzed (Participants) | 16 | 35 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.2 (1.0) | 4.2 (1.0) | 4.2 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 9 | 24 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 35 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 35 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Magnetic Resonance Imaging (MRI) Global Chest Score [Mean (Standard Deviation); unit: score on a scale] — MRI scans assessed semi-quantitatively via a standardized chest MRI scoring system. Each participant had 6 lobes scored using 7 scoring parameters:1)Bronchiectasis/wall thickening 2)Mucus plugging 3)Abscesses/sacculations 4)Consolidations 5)Special findings 6)Mosaic pattern 7)Perfusion abnormalities. For each of 7 parameter, there were scores of 6 lobes (score of each lobe :0=normal value, 1=<50 percent(%) of lobe involved and 2=>=50% of lobe involved). MRI global score was calculated as sum of parameters 1 to 7. MRI total score is ranged from 0-84. Higher score indicate more lobe involvement. Population: Baseline population included all randomized participants who have received at least 1 dose of study drug. Here "number analyzed" signifies participants who were evaluable for this outcome measure at the specified time point.
  score on a scale
    number analyzed (Participants) | 15 | 34 | 49
    (all) | 21.4 (9.3) | 17.6 (9.7) | 18.8 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Absolute Change From Baseline in MRI Global Chest Score at Week 48
Description: MRI scans assessed semi-quantitatively via a standardized chest MRI scoring system. Each participant had 6 lobes scored using 7 scoring parameters:1) Bronchiectasis/wall thickening 2) Mucus plugging 3) Abscesses/sacculations 4) Consolidations 5) Special findings 6)Mosaic pattern 7) Perfusion abnormalities. For each of 7 parameter, there were scores of 6 lobes (score of each lobe : 0= normal value, 1 = <50% of lobe involved and 2 = >=50% of lobe involved). MRI global score was calculated as sum of parameters 1 to 7. MRI total score is ranged from 0-84. Higher score indicate more lobe involvement.
Time Frame: From Baseline at Week 48
Population: Full Analysis Set (FAS) included all randomized participants who carried the intended CF transmembrane conductance regulator gene (CFTR) allele mutation and received at least 1 dose of study drug in Part 1. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part 1: LUM/IVA: Participants weighing <14 kg at screening received LUM 100 mg/IVA 125 mg FDC q12h in placebo-controlled period for 48 weeks. Participants weighing >=14 kg at screening received LUM 150 mg/IVA 188 mg FDC q12h in placebo-controlled period for 48 weeks.
Arm/Group | Part 1: Placebo | Part 1: LUM/IVA
Number analyzed (Participants) | 15 | 32
score on a scale | -0.3 (6.1) | -1.7 (6.6)
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: LUM/IVA; Test type: Superiority; Mean Difference = -1.5, 95% CI 2-sided [-5.5 to 2.6]

2. Secondary Outcome: Part 1: Absolute Change in Lung Clearance Index2.5 (LCI2.5) Through Week 48
Description: LCI2.5 represents the number of lung turnovers required to reduce the end-tidal inert gas concentration to 1/40th of its starting value.
Time Frame: From Baseline Through Week 48
Population: FAS.
Measure: Mean (95% Confidence Interval); unit: lung clearance index
Arm/Group | Part 1: Placebo | Part 1: LUM/IVA
Number analyzed (Participants) | 16 | 35
lung clearance index | 0.32 [-0.20 to 0.84] | -0.37 [-0.85 to 0.10]

3. Secondary Outcome: Part 1: Absolute Change in Weight-for-age Z-score at Week 48
Description: The z-score is a statistical measure to describe whether a value was above or below the standard. A z-score of 0 is equal to the standard. Lower numbers indicate values lower than the standard and higher numbers indicate values higher than the standard.
Time Frame: From Baseline at Week 48
Population: FAS.
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part 1: Placebo | Part 1: LUM/IVA
Number analyzed (Participants) | 16 | 35
z-score | -0.07 [-0.24 to 0.11] | 0.13 [-0.01 to 0.27]

4. Secondary Outcome: Part 1: Absolute Change in Stature-for-age Z-score at Week 48
Description: as for outcome 3
Time Frame: From Baseline at Week 48
Population: FAS.
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part 1: Placebo | Part 1: LUM/IVA
Number analyzed (Participants) | 16 | 35
z-score | 0.10 [-0.04 to 0.24] | 0.09 [-0.05 to 0.22]

5. Secondary Outcome: Part 1: Absolute Change in Body Mass Index (BMI)-For-age Z-score at Week 48
Description: BMI was defined as weight in kilogram (kg) divided by squared height in meters (m^2). The z-score is a statistical measure to describe whether a value was above or below the standard. A z-score of 0 is equal to the standard. Lower numbers indicate values lower than the standard and higher numbers indicate values higher than the standard.
Time Frame: From Baseline at Week 48
Population: FAS.
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part 1: Placebo | Part 1: LUM/IVA
Number analyzed (Participants) | 16 | 35
z-score | -0.24 [-0.55 to 0.07] | 0.20 [-0.02 to 0.41]

ADVERSE EVENTS:
Time Frame: From Day 1 up to Week 98 (Part 1: From Day 1 up to Week 48; Part 2: From Week 48 up to Week 98)
Description: MedDRA 23.1 applied for Part 1 and MedDRA 24.0 applied for Part 2.
Arm/Group | Part 1: Placebo | Part 1: LUM/IVA | Part 2: Overall LUM/IVA
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/35 | 0/49
Serious Adverse Events (participants affected / at risk) | 2/16 | 7/35 | 12/49
Other Adverse Events (participants affected / at risk) | 16/16 | 33/35 | 41/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=16) | Part 1: LUM/IVA (N=35) | Part 2: Overall LUM/IVA (N=49)
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 3 | 3
Otitis media (Infections and infestations) | 0 | 0 | 1
Pseudomonas bronchitis (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Sedation complication (Injury, poisoning and procedural complications) | 0 | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=16) | Part 1: LUM/IVA (N=35) | Part 2: Overall LUM/IVA (N=49)
Abdominal pain (Gastrointestinal disorders) | 2 | 7 | 6
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 3
Post-tussive vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 4
Pyrexia (General disorders) | 3 | 6 | 2
Bacterial disease carrier (Infections and infestations) | 2 | 0 | 3
Bronchitis (Infections and infestations) | 1 | 2 | 6
Conjunctivitis (Infections and infestations) | 1 | 1 | 1
Enterobiasis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 3 | 2
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 9 | 15 | 11
Nasopharyngitis (Infections and infestations) | 8 | 22 | 19
Otitis media (Infections and infestations) | 1 | 3 | 2
Rhinitis (Infections and infestations) | 6 | 9 | 8
Sinusitis (Infections and infestations) | 1 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 2
Viral infection (Infections and infestations) | 1 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 3
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2
Staphylococcus test positive (Investigations) | 1 | 1 | 3
Headache (Nervous system disorders) | 2 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0
Astigmatism (Eye disorders) | 0 | 2 | 1
Blepharospasm (Eye disorders) | 1 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 1
Faeces pale (Gastrointestinal disorders) | 2 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 2 | 0
Pseudomonas test positive (Investigations) | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT03625466/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT03625466/SAP_001.pdf